CLINICAL TRIAL: NCT03830528
Title: A Phase I Study of KW-6356 in Japanese and Caucasian Healthy Adults
Brief Title: A Study of Single and Multiple Doses of KW-6356 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6356-004
Record Dates: First submitted 2019-02-03; First posted 2019-02-05 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A-1 (Experimental): There will be 3 cohorts of Japanese healthy men dosed with single doses of KW-6356 (3 planned dose levels) or with placebo.
  Interventions: Drug: KW-6356 Low Dose
- Part A-2 (Experimental): There will be 3 cohorts of Japanese healthy men dosed with single doses of KW-6356 (3 planned dose levels) or with placebo.
  Interventions: Drug: KW-6356 Middle Dose
- Part A-3 (Experimental): There will be 3 cohorts of Japanese healthy men dosed with single doses of KW-6356 (3 planned dose levels) or with placebo.
  Interventions: Drug: KW-6356 High Dose
- Part B (Experimental): There will be one cohort of Japanese healthy men dosed with multiple doses of KW-6356 or placebo and one potential additional cohort (KW-6356 dose as determined in Part A or placebo)
  Interventions: Drug: KW-6356 X Dose
- Part C-1 (Experimental): There will be 2 cohort of Japanese and Caucasian healthy men dosed with multiple doses of KW-6356 (KW-6356 dose as determined in the previous studies)
  Interventions: Drug: KW-6356 Y Dose
- Part C-2 (Experimental): There will be 2 cohort of Japanese and Caucasian healthy men dosed with multiple doses of KW-6356 (KW-6356 dose as determined in the previous studies)
  Interventions: Drug: KW-6356 Y Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KW-6356 Low Dose — KW-6356 will be administered as single doses.
  Arms: Part A-1
Drug: KW-6356 Middle Dose — KW-6356 will be administered as single doses.
  Arms: Part A-2
Drug: KW-6356 High Dose — KW-6356 will be administered as single doses.
  Arms: Part A-3
Drug: KW-6356 X Dose — KW-6356 will be administered as multiple doses.
  Arms: Part B
Drug: KW-6356 Y Dose — KW-6356 will be administered for Japanese healthy men as multiple doses.
  Arms: Part C-1; Part C-2
Drug: Placebo — All study cohorts (except Part C) are placebo controlled.
  Arms: Placebo

SUMMARY:
Phase I study to assess the safety, tolerability and pharmacokinetics of single and multiple doses of KW-6356 in healthy volunteers

DETAILED DESCRIPTION:
The study will have 3 parts:

* In Part A and Part B, a placebo-controlled double-blind study will be conducted to investigate safety, tolerability and pharmacokinetics of a single dose and 14 days multiple doses of KW-6356 in Japanese healthy men, respectively
* In Part C, an open-label study will be conducted to investigate safety, tolerability and pharmacokinetics of 7 days multiple doses of KW-6356 in Japanese and Caucasian healthy men

ELIGIBILITY:
Inclusion Criteria:

* Individuals who provided freely-given written consent for participating in this study
* Men aged 20 ≥ and < 45 at the time of informed consent;

  * Japanese individuals without mixed marriage for at least last two generations, for participating Part A and Part B
  * Japanese and Caucasian individuals without mixed marriage for at least last two generations, for participating Part C
* Individuals with BMI ≥ 18.5 and < 30.0
* Individuals with screening results of; resting pulse rate: 40 to 100 bpm, systolic blood pressure: 91 to 140 mmHg, diastolic blood pressure: 40 to 90 mmHg

Exclusion Criteria:

* Individuals with any current diseases requiring treatment
* Individuals with current cerebrovascular, gastrointestinal, cardiovascular, hematologic, renal, or liver diseases
* Individuals with current symptomatic allergy
* Individuals with current or past drug allergy
* Individuals with current or past psychiatric disorders
* Individuals with a history of any autoimmune diseases or malignant tumor
* Individuals with alcohol or drug dependence, or those who showed any positive result(s) in drug abuse tests
* Individuals with a history of congestive heart failure, hypokalemia, hypocalcemia, or QT prolongation syndrome
* Individuals with positive result in any of viral infection tests (HBs antigen, HBs antibody, HBc antibody, HCV antibody, HIV antigen and antibody, and HTLV-1 antibody) or syphilis tests (RPR and TP antibody) at screening.
* Individuals with abnormality in standard 12-lead ECG that the investigator or subinvestigator determined as clinically significant at screening, Day -1, and before administration of the study drug on Day 1.
* Individuals who participated in clinical trial(s) of any medical products and received administration of those within 4 months prior to the study drug administration in the current study
* Individuals who used drugs (including non-prescription drugs, external preparation, vitamins, health supplements, and herbal medicines) within 2 weeks prior to the study drug administration
* Individuals who consumed grapefruit, or any food and beverage containing grapefruit or St John's Wort within 1 week prior to the study drug administration
* Individuals who smoked or used stop-smoking aid products (including chewing or eating nicotine-containing products, or application of nicotine patches) within 4 weeks prior to the study drug administration
* Individuals who admitted to the hospital or had surgery within 3 months prior to the study drug administration
* Individuals who had any of the following blood drawing for donation, clinical trial, or any other reasons prior to the study drug administration; ≥ 400 mL blood collection within 3 months; ≥ 200 mL blood collection within 4 weeks; or blood collection for pheresis (such as plasmapheresis or plateletpheresis) donation, clinical trial, or any other reasons within 2 weeks
* Individuals who did not agree to use appropriate contraceptive measures from the day of admission to 12 weeks after the last administration of study drug. The appropriate contraceptive measures are defined as refraining from sexual activity or combining two contraceptive methods including condom, oral contraceptives, intrauterine contraceptive devices or pessary.
* Any other individuals who were determined as not suitable for participating in this study by the investigator or subinvestigator

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Part A Number and percentage of subjects with treatment-emergent adverse events | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
Part B Number and percentage of subjects with treatment-emergent adverse events | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
Part C Profiles of pharmacokinetics of plasma KW-6356 concentrations | Starting about 24 hours before dosing and continued until about 7-14 days after last dose

SECONDARY OUTCOMES:
Part A Profiles of pharmacokinetics of plasma KW-6356 concentrations | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
Part B Profiles of pharmacokinetics of plasma KW-6356 concentrations | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
Part C Number and percentage of subjects with treatment-emergent adverse events | Starting about 24 hours before dosing and continued until about 7-14 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Co. LTA Sumida Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tayama T, Ishiuchi M, Sugiyama K, Oka Y, Maeda H, Nagata Y, Hruska M, Kagawa Y. Safety, Tolerability, and Pharmacokinetics of the Novel Adenosine A2A Antagonist/Inverse Agonist KW-6356 Following Single and Multiple Oral Administration in Healthy Volunteers. Clin Pharmacol Drug Dev. 2023 Aug;12(8):801-809. doi: 10.1002/cpdd.1222. Epub 2023 Jan 22. PMID 36683291